CLINICAL TRIAL: NCT06686823
Title: Effects of a Cognitive Training Program on Chemotherapy-induced Cognitive Impairment (Chemobrain) in Breast Cancer Patients Undergoing Active Treatment: A Randomized Controlled Trial
Brief Title: Effects of a Cognitive Training Program on Chemotherapy-induced Cognitive Impairment (Chemobrain) in Breast Cancer Patients Undergoing Active Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Prof. Dr. Eduardo J Fernández Rodríguez, Professor, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHEMOBRAIN MAMA
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Cancer-related Cognitive Impairment; Oncology; Breast Cancer; Cognitive Training; Everyday Cognition; Clinical Trials
Keywords: Cancer-related cognitive impairment; Oncology; Breast Cancer; Cognitive training; Clinical trials; Functional status
MeSH Terms: conditions — Neoplasms; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Education Program (Active Comparator): Instructions and recommendations will be provided in an informative leaflet to promote an active and healthy lifestyle, encouraging self-care and good practices. This leaflet will include the new WHO guidelines, which recommend specific measures to reduce the risk of cognitive decline. These measures are: Eating healthy foods, engaging in physical activity, maintaining social connections, playing challenging cognitive games, getting good sleep, managing stress, staying hydrated, and avoiding smoking and excessive alcohol consumption.
  Interventions: Behavioral: Health Education Program
- Cognitive Training Program (Experimental): The cognitive training program (CT) focused on everyday cognition (EC) will be conducted individually. Each participant will receive a dossier specifically designed for the study.
  The intervention will consist of four training periods over a duration of 4 months (Period 1, P1; Period 2, P2; Period 3, P3; Period 4, P4), with 20 activities each. Each period will last one month (5 activities per week).
  Interventions: Behavioral: Cognitive Training Program

INTERVENTIONS:
Behavioral: Health Education Program — n informative leaflet will promote a healthy lifestyle with WHO guidelines to reduce cognitive decline, recommending a balanced diet, physical activity, social engagement, cognitive games, good sleep, stress management, hydration, and avoiding smoking and excessive alcohol.
  Arms: Health Education Program
Behavioral: Cognitive Training Program — The cognitive training program (CT) on everyday cognition (EC) will be individualized, with each participant receiving a tailored dossier. The intervention includes four 1-month training periods (P1-P4), each featuring 20 activities, conducted at a rate of 5 activities per week over 4 months.
  Arms: Cognitive Training Program

SUMMARY:
Introduction: Given the increase in breast cancer survival rates, resulting from technological and biomedical advancements, it is essential to conduct an exhaustive study of the secondary symptoms associated with the oncological disease process. One of the most common and often underestimated symptoms is cancer-related cognitive impairment (CRCI).

Objective: To assess the effectiveness of a cognitive training program in managing CRCI in individuals with breast cancer undergoing active treatment.

Methodology: This is a randomized controlled clinical trial with two parallel groups: an Intervention Group (IG) and a Control Group (CG). The study population will consist of individuals with a new diagnosis of breast cancer. A required sample size of 50 participants has been estimated, with 25 in each group, to detect a difference equal to or greater than 2.95 points on the MoCA (Montreal Cognitive Assessment) questionnaire for cognitive impairment. All participants will receive an educational leaflet based on the new WHO guidelines, which recommend specific measures to reduce the risk of cognitive decline. In addition to this informative leaflet, the IG will receive a personalized cognitive training program (CT) focused on everyday cognition (EC). Each participant will be provided with a dossier containing 80 intervention sessions. The program will be divided into four training periods (P1-P4), each consisting of 20 activities, and each period will be conducted over one month. A baseline evaluation and a follow-up at 4 months post-intervention will be conducted for both groups. The assessments will measure sociodemographic and clinical variables, as well as study-related change variables related to cognitive impairment: Cognitive function (MoCA test), Everyday Cognition (PECC), Anxiety (Hamilton), Functionality (LB), Sleep quality (PSQI), Quality of life (ECOG), and Subjective memory complaints (FACT-COG).

Impact: The results of this study could lead to the design of specific cognitive interventions and the establishment of protocols for breast cancer patients undergoing active treatment. These interventions may help manage one of the most underestimated symptoms in this patient population, CRCI, whose incidence is increasing due to the higher survival rates in this disease.

DETAILED DESCRIPTION:
Introduction: Given the increase in breast cancer survival rates, resulting from technological and biomedical advancements, it is essential to conduct an exhaustive study of the secondary symptoms associated with the oncological disease process. One of the most common and often underestimated symptoms is cancer-related cognitive impairment (CRCI).

Objective: To assess the effectiveness of a cognitive training program in managing CRCI in individuals with breast cancer undergoing active treatment.

Methodology: This is a randomized controlled clinical trial with two parallel groups: an Intervention Group (IG) and a Control Group (CG). The study population will consist of individuals with a new diagnosis of breast cancer. A required sample size of 50 participants has been estimated, with 25 in each group, to detect a difference equal to or greater than 2.95 points on the MoCA (Montreal Cognitive Assessment) questionnaire for cognitive impairment. All participants will receive an educational leaflet based on the new WHO guidelines, which recommend specific measures to reduce the risk of cognitive decline. In addition to this informative leaflet, the IG will receive a personalized cognitive training program (CT) focused on everyday cognition (EC). Each participant will be provided with a dossier containing 80 intervention sessions. The program will be divided into four training periods (P1-P4), each consisting of 20 activities, and each period will be conducted over one month. A baseline evaluation and a follow-up at 4 months post-intervention will be conducted for both groups. The assessments will measure sociodemographic and clinical variables, as well as study-related change variables related to cognitive impairment: Cognitive function (MoCA test), Everyday Cognition (PECC), Anxiety (Hamilton), Functionality (LB), Sleep quality (PSQI), Quality of life (ECOG), and Subjective memory complaints (FACT-COG).

Ethical Considerations: The study will be conducted after obtaining approval from the Clinical Research Ethics Committee of the Salamanca Health Area. Informed consent will be obtained from all study participants, and data protection will be ensured.

Impact: The results of this study could lead to the design of specific cognitive interventions and the establishment of protocols for breast cancer patients undergoing active treatment. These interventions may help manage one of the most underestimated symptoms in this patient population, CRCI, whose incidence is increasing due to the higher survival rates in this disease.

ELIGIBILITY:
Inclusion Criteria:

Being an adult (18 years or older). Having a recent histopathological diagnosis of newly diagnosed breast cancer and starting oncological treatment.

Being fully capable of performing daily functions. Willingness to voluntarily participate in the study and signing the informed consent.

Exclusion Criteria:

Lack of literacy skills or significant language comprehension deficit. Diagnosis of a Central Nervous System tumor or participation in another cognitive stimulation program.

Clinical diagnosis of a neurocognitive disorder as defined in the DSM-V.

Withdrawal Criteria:

Dropping out of the program or not completing the final evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function | Baseline; "4 months final";
  The Montreal Cognitive Assessment Test (MoCA Test) Version 8.3. This test detects mild cognitive impairment (MCI) by assessing executive functions, attention, abstraction, memory, calculation, and orientation. It takes about 10 minutes to administer. The maximum score is 30 points, with scores below 26 indicating MCI.
Subjective Perception of Cognitive Impairment in Cancer Patients | Baseline; "4 months final";
  FACT-COG (Version 3) (24): This 37-item questionnaire is divided into six cognitive domains: memory, concentration, mental acuity, verbal fluency, functional interference, and multitasking ability. Additionally, it includes two subscales: "notability" (comments from others) and "perceived impact of cognitive impairment on quality of life." Respondents indicate the frequency of each occurrence over the past 7 days on a 5-point Likert scale, from 0 ("never") to 4 ("several times a day"). The scores from the individual subscales are summed to determine the total FACT-Cog score, ranging from 0 to 148, with higher scores indicating better cognitive functioning.

SECONDARY OUTCOMES:
Everyday Cognition | Baseline; "4 months final";
  Test for the Evaluation of Everyday Cognition (PECC) (18): This test measures an individual's ability to solve 12 real-life situations in areas such as medication management, administrative tasks, financial management, meal preparation, transportation, and shopping, thus assessing functional capacity in daily life. The administration time is 35 minutes.
Anxiety | Baseline; "4 months final";
  Hamilton Anxiety Rating Scale (19): A clinical assessment tool used to measure the level of anxiety experienced by a person. It consists of 14 items, each with five response options ranging from "not present" to "very severe." The final score can be 17 or less (mild anxiety), between 18 and 24 (moderate anxiety), and between 25 and 30 (severe anxiety).
Functionality | Baseline; "4 months final";
  Lawton and Brody Instrumental Activities of Daily Living (IADL) Scale (20): Designed to evaluate autonomy in instrumental activities in older adults. It takes about 4 minutes to administer, scoring each item as 0 or 1, with a total score of 8.
Sleep Quality | Baseline; "4 months final";
  Pittsburgh Sleep Quality Index (PSQI) (21): Designed to measure sleep quality in individuals aged 24 to 83 years. It takes 5-10 minutes to administer. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
Subjective Memory Failures | Baseline; "4 months final";
  Everyday Memory Failures Questionnaire (23): It includes categories such as "talking, reading, and writing," "names and faces," "actions," and "learning new things." Responses are given on a 9-point Likert scale, ranging from "Not at all in the last 3 months" to "More than once a day." Due to the complexity of the nine options, some authors use fewer response options.

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon request in the GREDOS scientific repository of the University of Salamanca once the study is completed. Link: https://gredos.usal.es/handle/10366/3823.
Supporting Information: Study Protocol, ICF, CSR
Access Criteria: The data will be available upon request in the GREDOS scientific repository of the University of Salamanca once the study is completed. Link: https://gredos.usal.es/handle/10366/3823.
URL: http://gredos.usal.es/